CLINICAL TRIAL: NCT00777582
Title: A Phase I, Randomised, 2 Period Cross Over Study to Determine the Comparative Bioavailability of Two Different Oral Formulations of AZD2281 in Cancer Patients With Advanced Solid Tumours
Brief Title: Phase I Comparative Bioavailability Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D0810C00024; 2008-003697-18 (EudraCT Number)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors
Keywords: Poly (ADP ribose) polymerases; Homologous Recombination Deficiency (HRD); Advanced solid tumours
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 300mg bid (twice daily) tablet dose
  Interventions: Drug: AZD2281
- Treatment B (Experimental): 400 mg twice daily (bid) capsule dose
  Interventions: Drug: AZD2281
- Treatment C (Experimental): 400mg bid (twice daily) tablet dose
  Interventions: Drug: AZD2281

INTERVENTIONS:
Drug: AZD2281 — Oral single dose formulation
  Other Names: Olaparib

SUMMARY:
The purpose of this phase I randomised cross over study is to determine and compare the bioavailability of two different oral formulations of AZD2281 in advanced solid tumour cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant advanced solid tumour, which is refractory to standard therapies (except Group 8 patients who must not be platinum refractory) or for which no suitable effective standard therapy exists
* Patients must have adequate organ and bone marrow function measured within 7 days prior to administration of study treatment
* Female patients must have evidence of non-child bearing status: negative urine or serum pregnancy test within 7 days of study treatment for women of child bearing, or postmenopausal status

Exclusion Criteria:

* Patients receiving chemotherapy, radiotherapy (except for palliative reasons) or any other anti-cancer therapy within 4 weeks of the last dose prior to study entry. Patients may continue the use of biphosphonates for bone metastases and corticosteroids
* Patients with symptomatic uncontrolled brain metastases
* Major surgery within 2 weeks of starting study and patients must have recovered from any effects of any major surgery
* Patients who are platinum refractory (Group 8 only)
* Patients with myelodysplastic syndrome/acute myeloid leukaemia (Group 8 only).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-10-27 (Actual); Primary Completion 2009-02-06 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PK Phase Primary Outcome: To determine the comparative bioavailability of a new tablet formulation of AZD2281 compared to the existing capsule formulation | Blood samples (12) will be taken at pre-defined intervals following dosing of a single capsule and a single tablet dose
Continued Supply Phase: To enable patients to continue to receive treatment with AZD2281. Safety and tolerability data will be collected to further determine the safety and tolerability of the capsule formulation of AZD2281 in these patients | every 28 days
Continued Supply Expansion Phase: To compare the safety and tolerability of the tablet and capsule formulation of AZD2281 in all patients: Safety, AEs, Physical Exam, vital signs | at every visit
Dose Escalation Phase of continued supply expansion: To determine safety & tolerability of higher than 200mg bid (to 400mg) of tablet & compare safety & tolerability profile of tablet with 400mg capsule | at every visit
Randomised tablet formulation continued supply expansion phase (Group 8): To determine the safety and tolerability profile of selected tablet dose schedules of the melt-extrusion (tablet) formulation. | at every visit

SECONDARY OUTCOMES:
PK Phase Secondary Outcome: To generate single dose PK data for the new tablet formulation in man, and to generate information on dose linearity for the new tablet formulation | Blood samples (12) will be taken at pre-defined intervals prior to and following dosing of a single capsule and a single tablet dose
To compare the extent of PARP inhibition achieved in peripheral blood mononuclear cells (PBMCs) following dosing of both the new tablet formulation and existing capsule formulation | Blood samples (4) will be taken at pre-defined intervals prior to and following dosing of a single capsule and a single tablet dose
To determine the safety and tolerability of AZD2281 for both the new tablet formulation and existing capsule formulations | every 28 days
Continued Supply Expansion Phase: To compare the steady state exposure achieved with 200mg bid tablet formulation and 400mg bid capsule formulation | at visit 3 and visit 4
Continued Supply Expansion Phase: To describe the efficacy data observed in patients treated with the capsule and the tablet | RECIST, Progression Free Survival, Best overall response and CA-125 response
Dose Escalation Phase of the continued supply expansion: To determine the single dose and steady state exposures achieved with higher doses of AZD2281 tablet formulation | at every visit
Dose Escalation Phase of the continued supply expansion: To compare between patients the single dose and steady state exposures of AZD2281 achieved with selected tablet doses and the 400mg bid capsule dose | at every visit
Dose Escalation Phase of the continued supply expansion: To describe the efficacy data observed in patients treated with the capsule formulation and the tablet formulation | at every visit
Randomised tablet formulation continued supply expansion phase (Group 8): To determine the single dose and steady state exposures achieved with the selected table dose schedules of AZD2281 melt-extrusion (tablet) formulation | at every visit
Randomised tablet formulation continued supply expansion phase (Group 8): To obtain a preliminary assessment of the effect of food on the exposure to AZD2281 following dosing of the melt-extrusion (tablet) formulation. | at every visit
Randomised tablet formulation continued supply expansion phase (Group 8): To describe the efficacy data observed in patients treated with the melt-extrusion (tablet) formulation | at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Stan Kaye, Professor, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (10):
- Research Site, Randwick, Australia
- Research Site, Leuven, Belgium
- Research Site, Bellinzona, Switzerland
- United Kingdom (7):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Northwood
  - Research Site, Oxford
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Mateo J, Moreno V, Gupta A, Kaye SB, Dean E, Middleton MR, Friedlander M, Gourley C, Plummer R, Rustin G, Sessa C, Leunen K, Ledermann J, Swaisland H, Fielding A, Bannister W, Nicum S, Molife LR. An Adaptive Study to Determine the Optimal Dose of the Tablet Formulation of the PARP Inhibitor Olaparib. Target Oncol. 2016 Jun;11(3):401-15. doi: 10.1007/s11523-016-0435-8. PMID 27169564
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Ang JE, Gourley C, Powell CB, High H, Shapira-Frommer R, Castonguay V, De Greve J, Atkinson T, Yap TA, Sandhu S, Banerjee S, Chen LM, Friedlander ML, Kaufman B, Oza AM, Matulonis U, Barber LJ, Kozarewa I, Fenwick K, Assiotis I, Campbell J, Chen L, de Bono JS, Gore ME, Lord CJ, Ashworth A, Kaye SB. Efficacy of chemotherapy in BRCA1/2 mutation carrier ovarian cancer in the setting of PARP inhibitor resistance: a multi-institutional study. Clin Cancer Res. 2013 Oct 1;19(19):5485-93. doi: 10.1158/1078-0432.CCR-13-1262. Epub 2013 Aug 6. PMID 23922302
- [Derived] Sandhu SK, Omlin A, Hylands L, Miranda S, Barber LJ, Riisnaes R, Reid AH, Attard G, Chen L, Kozarewa I, Gevensleben H, Campbell J, Fenwick K, Assiotis I, Olmos D, Yap TA, Fong P, Tunariu N, Koh D, Molife LR, Kaye S, Lord CJ, Ashworth A, de Bono J. Poly (ADP-ribose) polymerase (PARP) inhibitors for the treatment of advanced germline BRCA2 mutant prostate cancer. Ann Oncol. 2013 May;24(5):1416-8. doi: 10.1093/annonc/mdt074. Epub 2013 Mar 22. No abstract available. PMID 23524863
- See also: D0810C00024_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1676&filename=D0810C00024_Study_Synopsis.pdf